CLINICAL TRIAL: NCT00829855
Title: Echocardiographic Evaluation of Hypertensive Acute Pulmonary Edema
Status: Completed | Type: Observational
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Collaborators: Ministry of Education, Research, Youth and Sport, Romania (Other)
Responsible Party: Principal Investigator, Mircea Cinteza, Professor, Carol Davila University of Medicine and Pharmacy
Other Study IDs: IDEI_242_2007; ID_216/PNII_242_2007
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Pulmonary Edema; Hypertension
Keywords: pulmonary edema; hypertension; echocardiography
MeSH Terms: conditions — Pulmonary Edema; Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients with hypertensive (systolic blood pressure ≥160 mmHg) acute pulmonary edema, evaluated within 120 minutes after admittance.
- 2: The same patients from group 1 followed-up at 48 to 96 hours.

SUMMARY:
Acute cardiogenic pulmonary edema (ACPE), one of the most severe forms of acute heart failure, represents 5% of hospital admissions. One of the most frequent phenomena encountered during ACPE is hypertensive crisis (hypertensive ACPE) but the mechanisms and causes of hypertensive ACPE are insufficiently understood. Few studies have evaluated the cardiac function during hypertensive ACPE, and these studies used only conventional echocardiography methods. New methods of evaluation of cardiac function in hypertensive ACPE (such as Tissue Doppler imaging) have not been used.

The objectives of this study are to evaluate presence and role of the following potential mechanisms of hypertensive ACPE: 1. acute myocardial dysfunction (systolic and diastolic); 2. silent transient myocardial ischemia; 3. acute mechanical left ventricular dyssynchrony; 4. dynamic mitral regurgitation; 5. inter-ventricular interaction. Conventional and Tissue Doppler echocardiography will be used to assess cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* acute onset of dyspnea within the preceding 8 hours
* respiratory distress and pulmonary rales at any level
* pulmonary congestion confirmed by chest radiography
* systolic blood pressure > 160 mmHg before treatment
* sinus rhythm
* signed informed consent

Exclusion criteria:

* acute myocardial infarction confirmed by myocardial necrosis markers (either CKMB or troponin I). Angina pectoris alone will not be excluded
* significant left sided valvular disease (more than moderate). Mitral regurgitation of any severity will not be excluded, due to the hypothesis of the role of dynamic mitral regurgitation in the pathogenesis of acute hypertensive pulmonary edema
* congenital heart disease
* cardiac tamponade
* rhythm and conduction disturbances that may have precipitated pulmonary edema, like sustained ventricular tachycardia and complete heart block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in the Cardiac Care Unit of an University and Emergency Hospital, with a diagnosis of acute cardiogenic pulmonary edema associated with hypertension (systolic blood pressure ≥160 mmHg)
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
acute myocardial dysfunction (systolic and diastolic) and/or dyssynchrony | acute event and 48 to 96 h after the event

SECONDARY OUTCOMES:
surrogate markers of silent transient myocardial ischemia | acute event and 48 to 96 h after the event
dynamic mitral regurgitation | acute event and 48 to 96 h after the event
inter-ventricular interaction | acute event and 48 to 96h after the event

CONTACTS AND LOCATIONS:
Overall Officials: Mircea Cinteza, MD, PhD, Principal Investigator — University of Medicine and Pharmacy "Carol Davila" Bucharest; Dragos Vinereanu, MD, PhD, Principal Investigator — University of Medicine and Pharmacy "Carol Davila" Bucharest; Andrei D Margulescu, MD, Study Chair — University of Medicine and Pharmacy "Carol Davila" Bucharest
Locations (1):
- Department of Cardiology, University and Emergency Hospital of Bucharest, Bucharest, Romania